CLINICAL TRIAL: NCT07062822
Title: The Role of Resisted Exercise and Kinesiology-Taping in Managing Knee Osteoarthritis in Overweight and Obese Individuals.
Brief Title: Resisted Exercise and Kinesiology-Taping in Managing Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Rec-01014 Jeyad Khan
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Resisted exercises
  Interventions: Other: Resisted exercise
- Group B (Placebo Comparator): kinesio-tapping
  Interventions: Other: kinesiology tapping

INTERVENTIONS:
Other: Resisted exercise — Patients in this group will be applied Kinesio taping 3 times per week over the study period of 6 weeks. Before the kinesio taping, the skin surface will be clean. Patients will positioned lying on their side, hip extended, and knee joint at 60° of flexion. The knee will be tape with an I-shaped kinesio tape starting at the origin of the rectus femoris, and a Y-shaped kinesio tape proximal to the superior patellar border. The taping will be no tension at its base, whereas the portion between the anchor and the superior patella will be stretched ≈40%.
  Arms: Group A
Other: kinesiology tapping — kinesiology tapping
  Arms: Group B

SUMMARY:
The study aims the Role of Resisted Exercise and Kinesiology Taping in Managing Knee Osteoarthritis in Overweight and Obese Individuals.

DETAILED DESCRIPTION:
The study focuses on understanding Knee osteoarthritis (OA) is a chronic progressive disease commonly seen in the elderly.The main symptoms include pain, joint stiffness, reduction in the range of motion (ROM), Crepitus during activity, inflammation and swelling. Furthermore, patients with knee OAMay suffer from joint deformity, muscle atrophy of the lower extremities, abnormal gait, orEven ambulatory inability As the quality of life of knee OA patients remains very poor,The pain reduction, muscle strength enhancement, deformity prevention, and function Improvement of knee OA are important issues in the aging population nee Osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a clinical diagnosis of knee osteoarthritis, confirmed by imaging (e.g., X-ray, MRI) or a physician's diagnosis based on clinical evaluation. This ensures that participants actually have the condition being studied.
* Pain Level: Moderate pain (e.g., 3-6 on the Visual Analog Scale or VAS): Participants should experience moderate pain levels during activities of daily living (ADLs), such as walking, climbing stairs, or squatting. This level of pain should be sufficient to demonstrate the potential effects of the interventions (resisted exercise and kinesiotaping).
* Impairments related to knee pain, such as difficulty walking, bending, or climbing stairs
* Stable Medical Condition: Participants should have stable health with no significant comorbidities (e.g., uncontrolled cardiovascular diseases, severe arthritis in other joints, or neurological disorders)

Exclusion Criteria:

* Severe Knee Deformities or Structural Damage: Individuals with severe joint deformities or advanced OA (e.g., bone-on-bone contact as observed on radiographs) may be excluded, as they may not respond to conservative interventions like resisted exercise or kinesiotaping
* Recent Knee Surgery: Exclude participants who have undergone knee surgery (e.g., total knee replacement, arthroscopy) within the past 6-12 months, as recovery from surgery may confound the results of the study.
* Other Inflammatory Joint Disorders: Participants with other inflammatory joint diseases (e.g., rheumatoid arthritis, gout, or psoriatic arthritis) should be excluded to ensure that the results are specifically related to knee OA, not other conditions that affect the joints.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-17 (Estimated); Primary Completion 2026-05-13 (Estimated); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 3 weeks
  A 10 cm horizontal line with "No Pain" (0) on the left and "Worst Pain" (10) on the right.

CONTACTS AND LOCATIONS:
Overall Officials: Ataur Rahman, MS-PT (CPPT), Principal Investigator — Riphah International University

IPD SHARING:
Plan to Share IPD: No